CLINICAL TRIAL: NCT05938686
Title: Home_Based Digital Mindful Dance Program for Breast Cancer Cases: Feasibility, Body-Mind Awareness and Quality of Life
Brief Title: Home_Based Digital Mindful Dance Program for Breast Cancer Cases
Acronym: Dance4BC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, I-Ching Hou, Associate Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NYCU112051AEF
Record Dates: First submitted 2023-06-29; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer; Quality of Life
Keywords: breast cancer; mindfulness; dance; home based digitalization; quality of life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Experimental): Home_Based Digital Mindful Dance Program for 12 weeks
  Interventions: Other: Home_Based Digital Mindful Dance Program
- Control Group (No Intervention): Routine care for 12 weeks.

INTERVENTIONS:
Other: Home_Based Digital Mindful Dance Program — Home_Based Digital Mindful Dance Program including warm up, dance and cool down for 60 minute with 12 weeks.
  Arms: Interventional Group

SUMMARY:
During COVID-19, telecare replaces face-to-face contact to maintain social distance and reduce the spread of the virus. The current epidemic is coming to the end. However, for breast cancer cases, no matter in the treatment or survival stage, they face physical and mental symptoms, such as "social isolation", which affects their quality of life. Studies have shown that mindfulness and dance can help breast cancer cases improve depression and quality of life, but most of them are conducted face-to-face. Online mindful/dance helped breast cancer cases without the limitations of the time, space, distance, and treatment status, but lacking enough evidence. The purpose of this study will to design a "home based digital mindful dance program" suitable for our breast cancer cases, and conduct clinical trial on its feasibility, mind and body awareness, and quality of life. Finally, through in-depth interviews, we will understand the subjective experience of breast cancer cases on the program. The research results are expected to provide an empirical reference for multi-care for breast cancer to our country and abroad.

DETAILED DESCRIPTION:
Since the outbreak of the COVID-19 global pandemic at the end of 2019, maintaining social distance has become an important strategy to avoid virus infection. Various interventional care intervention that traditionally need to be implemented face-to-face also urgently need to be adjusted to online with the assistance of digital technology tools. Provide (e.g. video clinic).

Although the current epidemic situation has tended to stabilize, however, for breast cancer patients, they are often in a state of "social isolation" physically and mentally from the beginning of diagnosis and treatment to the survival stage after treatment.

Because breast cancer patients often need to receive chemotherapy, they are affected by drugs and produce bone marrow suppression, resulting in lower autoimmune function than normal people. They belong to a high-risk group of infection, and they need to take self-protection measures and reduce going to public places. Even if all cancer treatments have been completed and are in the survival period, some patients may choose to leave the hard-working workplace early due to fear of cancer recurrence or social prejudice to reduce stress and health threats, but they are also worried about the burden on their families and loss of life. Center of gravity, when multiple psychological pressures continue to accumulate, it is easy to cause emotional distress such as anxiety or depression, and it also seriously affects interpersonal relationships and social skills. Therefore, whether it is in the treatment stage or the survival stage, the body and mind often suffer from a negative state like "social isolation" .

Mindfulness is consciously aware of the present body, mind and environment, and maintains an objective, permissive, and non-judgmental attitude. Its exercises include breathing observation, body scanning, meditation, walking, yoga, and relaxation techniques. Dance is a dual-task activity that integrates cognitive, motor, and emotional tasks through a combination of spatial awareness, motor coordination, balance, endurance, and interaction. Past studies have pointed out that mindful dance measures through mindfulness techniques, dance movements, or a combination of the two can help breast cancer patients improve their quality of life, reduce depression, anxiety, pain, fatigue symptoms, improve sleep quality, and reduce the fear of cancer recurrence and many other benefits.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer with any stage and any treatment status

Exclusion Criteria:

* mental illness

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — more than 20 years old
Enrollment: 104 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Baseline EORTC QLQ-C30 | Baseline
  Baseline Taiwan Chinese version of the European Organisation for Research and Treatment of Cancer Quality of Life - Core 30 (version 3). The minimum and maximum values are 0 and 100, and higher scores mean a better outcome.
Change of EORTC QLQ-C30 at 12th week | 12th week
  Change from baseline Taiwan Chinese version of the European Organisation for Research and Treatment of Cancer Quality of Life - Core 30 (version 3) to 12th week. The minimum and maximum values are 0 and 100, and higher scores mean a better outcome.
Baseline QLQ-BR23 | Basline
  Baseline Taiwan Chinese version of the European Organisation for Research and Treatment of Cancer Quality of Life - Breast 23 (version 3). The minimum and maximum values are 0 and 100, and higher scores mean a better outcome.
Change of QLQ-BR23 at 12th week | 12th week
  Change from baseline Taiwan Chinese version of the European Organisation for Research and Treatment of Cancer Quality of Life - Breast 23 (version 3) to 12th week. The minimum and maximum values are 0 and 100, and higher scores mean a better outcome.
Baseline Mindful Attention Awareness Scale | Basline
  Baseline Mindful Attention Awareness Scale. Based on a mean of all items, MAAS scores can range from 1 to 6. Higher scores indicate greater mindfulness
Change of Mindful Attention Awareness Scale at 12th week | 12th week
  Change from baseline Mindful Attention Awareness Scale to 12th week. Based on a mean of all items, MAAS scores can range from 1 to 6. Higher scores indicate greater mindfulness

SECONDARY OUTCOMES:
Baseline Physical Activity Scale | Basline
  Baseline Physical Activity Scale. The minimum and maximum values are 1 and 4, and higher scores mean a better physical activity.
Change of Physical Activity Scale at 12th week | 12th week
  Change from baseline Physical Activity Scale to 12th week. The minimum and maximum values are 1 and 4, and higher scores mean a better outcome.
Feasibility Test at 12th week | 12th week
  Feasibility Test at 12th week.The minimum and maximum values are 1 and 4, and higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: I-Ching Hou, PhD, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang-Ming University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No